CLINICAL TRIAL: NCT05126381
Title: Population Pharmacokinetic - Pharmacodynamic Models of Chronic Disease Therapeutics for Smokers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021LCYJ040
Record Dates: First submitted 2021-11-02; First posted 2021-11-19 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2022-12

CONDITIONS: Chronic Disease; Smoking
Keywords: Population Pharmacokinetics/ Pharmacodynamics; Gene polymorphism; Smoking
MeSH Terms: conditions — Chronic Disease; Smoking | interventions — Smoking Devices

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Smoker with taking levamlodipine besylate tablets: The subjects are allowed to smoke during the time taking levamlodipine besylate tablets.
  Interventions: Behavioral: Smoking
- Non-smoker with taking levamlodipine besylate tablets: The subjects are not allowed to smoke during the time taking levamlodipine besylate tablets.
  Interventions: Behavioral: non-somking
- Smoker with taking metformin sustained-release tablets: The subjects are allowed to smoke during the time taking metformin sustained-release tablets。
  Interventions: Behavioral: Smoking
- Non-smoker with taking metformin sustained-release tablets: The subjects are not allowed to smoke during the time taking metformin sustained-release tablets.
  Interventions: Behavioral: non-somking

INTERVENTIONS:
Behavioral: Smoking — The Study contains patients who are allowed to smoke
  Groups: Smoker with taking levamlodipine besylate tablets; Smoker with taking metformin sustained-release tablets
Behavioral: non-somking — The Study contains patients who are not allowed to smoke
  Groups: Non-smoker with taking levamlodipine besylate tablets; Non-smoker with taking metformin sustained-release tablets

SUMMARY:
Purpose of study: Establishing population pharmacokinetic - pharmacodynamic models of chronic disease therapeutics for smoking patients to investigate the effects of gender, age, body weight, liver function, kidney function, nicotine, polycyclic aromatic hydrocarbon related metabolic enzymes and drug related metabolic enzymes gene polymorphism on steady-state drug concentration and efficacy in chronic smoking patients after taking drugs.

Object of study: Smoking and non-smoking patients taking levamlodipine besylate tablets or metformin sustained-release tablets.

DETAILED DESCRIPTION:
Purpose of study: Establishing population pharmacokinetic - pharmacodynamic modes of chronic disease therapeutics for smoking patients to investigate the effects of gender, age, body weight, liver function, kidney function, nicotine, polycyclic aromatic hydrocarbon related metabolic enzymes and drug related metabolic enzymes gene polymorphism on steady-state drug concentration and efficacy in chronic smoking patients after taking drugs.

Object of study: Smoking and non-smoking patients taking Levamlodipine besylate tablets or metformin sustained-release tablets.

Parameters of study： PK parameters: drug plasma concentration. PD parameters: blood pressure or blood sugar. covariates: Gender, age, height, weight, BMI, liver function (ALT, AST, TP, TBIL), kidney function (Scr, UA, UREA), nicotine plasma concentration, cigarette related metabolic enzyme gene (CYP1A1, CYP1A2) polymorphism and drug-related metabolic enzyme gene (CYP3A4, CYP3A5, MATE1), MARE2, OCT2) polymorphism, etc.

Safety : adverse events occurred during the test.

ELIGIBILITY:
Inclusion Criteria:

According to the selection criteria for non-smokers:

No previous smoking history;Or previous smokers who had quit smoking for more than 6 months prior to enrollment.

A smoker joins the queue by:

1. Have smoked for more than one year (more than one cigarette per day on average and more than six months continuously) and have not quit at present.
2. Agree to smoke cigarettes sold in the market according to the requirements of the program.

Both smokers and non-smokers were forced to meet additional inclusion criteria at the cost of a smoker:

1. Age: 18-70 (boundary value included), no gender limitation;
2. Patients who meet one of the following conditions:

   ① Patients who were previously diagnosed with hypertension, were taking levamlodipine besylate tablets for antihypertensive therapy, and were managed according to hypertensive lifestyle (diet and exercise) for a long time.

   ② Patients who were previously diagnosed with type 2 diabetes, were taking metformin sustained-release tablets for hypoglycemic treatment, and were managed according to diabetic lifestyle (diet and exercise) for a long time.
3. Fixed dosing regimen was used one month before enrollment, and the regimen could be continued after enrollment.
4. Subjects understand the risks and regulations of the study and can abide by the study protocol, voluntarily participate in the study and sign the informed consent.

Exclusion Criteria:

1. Have a history of alcohol abuse (drinking more than 14 units of alcohol per week, 1 unit =350 mL beer or 44 mL 40% alcohol spirits or 150 mL wine) or have a history of alcohol abuse and have been abstinent for less than 3 months.
2. The subject has a history of pathophysiological conditions affecting drug absorption (such as inability to swallow, vomiting, diarrhea, etc.) or gastrointestinal surgery affecting drug absorption.
3. HBsAg, HCV or syphilis antibody tested positive in the past.
4. Pregnant and lactating women.
5. The investigator considers that the subjects are not suitable to participate in this study due to safety or compliance factors.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects were mainly selected for outpatient follow-up
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-01-13 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Drug plasma steady state concentrations | Blood samples were collected 30 minutes before administration
  drug plasma steady state concentrations are regard as the PK parameters

OTHER OUTCOMES:
Blood pressure levels | Blood pressure levels were collected 30 minutes before administration
  Blood pressure levels are regard as the PD parameters
Blood glucose levels | Blood glucose levels were collected 30 minutes before administration
  Blood glucose levels are regard as the PD parameters

CONTACTS AND LOCATIONS:
Overall Officials: Yu Xian, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- Yu Xian, Chongqing, China

IPD SHARING:
Plan to Share IPD: No